CLINICAL TRIAL: NCT04139746
Title: Pneumatic Retinopexy Preceded by Drainage of Subretinal Fluid for the Treatment of Severe Bullous Retinal Detachment
Brief Title: Pneumatic Retinopexy for Severe Bullous Retinal Detachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Francesco Semeraro, Prof. Francesco Semeraro, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitreo004
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Retina Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Scleral Buckling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scleral Buckling (Active Comparator): Scleral Buckling represents the gold standard for retinal detachment in young phakic patients.
  Interventions: Procedure: Scleral Buckling
- Drainage-Injection-Pneumoretinopexy (Experimental): Drainage-Injection-Pneumoretinopexy is a modified pneumatic retinopexy technique, in which, before injecting the gas, the drainage of the subretinal fluid is performed with a simultaneous injection of balanced salt solution (BSS) in the vitreous chamber.
  Interventions: Procedure: Drainage-Injection-Pneumoretinopexy

INTERVENTIONS:
Procedure: Scleral Buckling — Limbal 360 degrees peritomy of the conjunctiva was performed and the four recti muscles were isolated with 4 silk threads 4-0. A width-2 mm silicone encircling band was placed and sutured with 5-0 mersilene on the 4 quadrants of the sclera. Anterior chamber paracentesis was performed, draining about 0.3 mL of aqueous humour, and a buckle (220, 501, 506, or 516; Mira, Waltham, MA, USA) was sutured over the break. In all cases, the drainage puncture was executed at a distance of 11 mm from the limbus, in the area of greatest amount of subretinal fluid. Soon after the drainage puncture, a balanced salt solution (BSS) injection was performed in order to compensate the escape of the subretinal fluid.
  Arms: Scleral Buckling
Procedure: Drainage-Injection-Pneumoretinopexy — According to the location of the sub-retinal fluid, a quadrant-flap of conjunctiva was opened. Indirect ophthalmoscopy evaluation was also used intraoperatively to localize the break and the subretinal fluid drainage site: in this area a vicryl 6-0 thread was passed through the sclera, about 9-10 mm posteriorly from the limbus, to facilitate the surgical maneuvers. The drainage puncture was performed 11 mm posteriorly from the limbus, having attention not to perform it directly above the site of the retinal break. In detail, a 2 mm radial sclera incision was created with a 15° disposable knife. The incision was cautiously deepened down to the choroid, which was finally perforated by a lachrymal dilator having a blunt tip. Soon after beginning the subretinal fluid drainage, an injection of BSS was performed in the opposite quadrant of the sclera (4 mm from the limbus) in order to allow an optimal spillage of the subretinal fluid and to flatten the retina.
  Arms: Drainage-Injection-Pneumoretinopexy

SUMMARY:
To compare the efficacy and safety outcomes of scleral buckling (SB) and drainage-injection-pneumoretinopexy (DIP), a modified pneumatic retinopexy technique, in which, before injecting the gas, the drainage of the subretinal fluid is performed with a simultaneous injection of balanced salt solution (BSS) in the vitreous chamber, for the treatment of severe superior bullous rhegmatogenous retinal detachment (SBRD).

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent;
* phakic patients aged < 60 years with no or minimal media opacity;
* single or multiple retinal breaks (within 1 clock hour) between 8 to 4 o'clock hours;
* patients' capability to maintain suggested head positioning for 5 days after the procedure.

Exclusion Criteria:

* retinal detachment with poor subretinal fluid (absence of severe SBRD);
* holes, lattice degeneration or traction within the inferior 4 clock hours;
* posterior retinal break, situated behind the equator, not suitable for cryotherapy;
* any sign of PVR or severe glaucoma;
* myopia above 10 diopters.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Anatomical reattachment of the retina | 12-month

SECONDARY OUTCOMES:
Refractive error change | 12-month

CONTACTS AND LOCATIONS:
Locations (1):
- Spedali Civili di Brescia, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No